CLINICAL TRIAL: NCT01752894
Title: DETErmination of the Duration of the Dual Antiplatelet Therapy by the Degree of the Coverage of The Struts on Optical Coherence Tomography From the Randomized Comparison Between Everolimus-eluting Stents(EES) Versus Biolimus A9-eluting Stents(BES)
Acronym: DETECT-OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2012-0047
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Angio guided PCI (Active Comparator)
  Interventions: Device: Angio-guided PCI with EES or BES
- OCT-guided PCI (Experimental)
  Interventions: Device: OCT-guided PCI with EES or BES
- BES (Active Comparator)
  Interventions: Device: PCI with BES under angio-guide or OCT guide
- EES (Experimental)
  Interventions: Device: PCI with EES under angio-guide or OCT guide
- Keep dual antiplatelet therapy (DAPT) (Active Comparator): Study subjects will be allocated into this arm with non-randomization method
  Interventions: Drug: Keep DAPT
- Discontinue Dual antiplatelet therapy (DAPT) (Active Comparator): Study subjects will be allocated into this arm with non-randomization method
  Interventions: Drug: Discontinue DAPT

INTERVENTIONS:
Device: Angio-guided PCI with EES or BES — Angio-guided intervention
  Arms: Angio guided PCI
Device: OCT-guided PCI with EES or BES — OCT-guided intervention
  Arms: OCT-guided PCI
Device: PCI with BES under angio-guide or OCT guide — biolimus A9-eluting stent.
  Arms: BES
Device: PCI with EES under angio-guide or OCT guide — everolimus eluting stent.
  Arms: EES
Drug: Keep DAPT — maintain DAPT for 12 months according to level of uncovered strut (>6%) at 3months OCT follow up after stent implantation.
  Arms: Keep dual antiplatelet therapy (DAPT)
Drug: Discontinue DAPT — discontinue DAPT according to level of uncovered strut (≤6%) at 3months OCT follow up after stent implantation.
  Arms: Discontinue Dual antiplatelet therapy (DAPT)

SUMMARY:
The purpose of the study is 1> to compare neointimal stent coverage after OCT-guided vs. Angio-guided PCI, 2> to compare neointimal stent coverage at 3 months after EES vs BES implantation, 3> to determine the duration of dual antiplatelet therapy by OCT measurement at 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 20 years old
* Patients with ischemic heart disease who are considered for coronary revascularization with stent implantation.
* Significant coronary de novo lesion (stenosis > 70% by quantitative angiographic analysis) treated by single DES ≤ 25mm
* Reference vessel diameter of 2.5 to 3.5 mm by operator assessment

Exclusion Criteria:

* Complex lesion morphologies such as aorta-ostial, unprotected left main, chronic total occlusion, graft, thrombosis, and restenosis
* Reference vessel diameter < 2.5 mm or > 4.0mm
* Heavy calcified lesions (definite calcified lesions on angiogram)
* Primary PCI for STEMI
* Contraindication to anti-platelet agents
* Treated with any DES within 3 months at other vessel
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2013-01-02; Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
percentage of neointimal coverage at 3 month-OCT after stent implantation | at 3 month-OCT after stent implantation

SECONDARY OUTCOMES:
The occurrence of the composite of cardiac death, MI, definite or probable stent thrombosis, and TIMI-defined major bleeding for 12 months | 12 months after PCI
percentage of malposition strut at 3 month-OCT after stent implantation | 3 months after PCI
The occurrence of the composite of All cause death, spontaneous MI, Target vessel revascularization and stroke. | 12 months after PCI
Target vessel revascularization | 12 months after PCI
TIMI-defined major bleeding for 12 months | 12 months after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jin IT, Kim Y, Heo SJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Cho DK, Ko YG, Choi D, Hong MK, Kim BK. Comparison of Short-term and Standard Duration Dual Antiplatelet Therapy in Elderly Patients: A Pooled Analysis of Five Korean Randomized Clinical Trials. Korean Circ J. 2025 Dec;55(12):1125-1137. doi: 10.4070/kcj.2025.0093. Epub 2025 Jul 14. PMID 41044734
- [Derived] Lee SY, Ahn CM, Yoon HJ, Hur SH, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. Early Follow-Up Optical Coherence Tomographic Findings of Significant Drug-Eluting Stent Malapposition. Circ Cardiovasc Interv. 2018 Dec;11(12):e007192. doi: 10.1161/CIRCINTERVENTIONS.118.007192. PMID 30562088
- [Derived] Lee SY, Kim JS, Yoon HJ, Hur SH, Lee SG, Kim JW, Hong YJ, Kim KS, Choi SY, Shin DH, Nam CM, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. Early Strut Coverage in Patients Receiving Drug-Eluting Stents and its Implications for Dual Antiplatelet Therapy: A Randomized Trial. JACC Cardiovasc Imaging. 2018 Dec;11(12):1810-1819. doi: 10.1016/j.jcmg.2017.12.014. Epub 2018 Feb 14. PMID 29454763